CLINICAL TRIAL: NCT01694966
Title: The Safety and Efficacy of Methylene Blue MMX® Modified Release Tablets Administered to Subjects Undergoing Screening or Surveillance Colonoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cosmo Technologies Ltd (Industry)
Responsible Party: Sponsor
Organization: CosmoTech (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: CB-17-01/06; 2012-003983-32 (EudraCT Number)
Record Dates: First submitted 2012-09-25; First posted 2012-09-27 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Methylene Blue MMX® 200mg (Active Comparator): Oral dose, 8 Methylene Blue MMX® tablets over a 4hr schedule
  Interventions: Drug: Methylene Blue MMX®
- Methylene Blue MMX® 100mg (Active Comparator): Oral dose, 4 Methylene Blue MMX® tablets and 4 Placebo tablets over a 4hr schedule
  Interventions: Drug: Methylene Blue MMX®; Drug: Placebo
- Placebo (Placebo Comparator): Oral dose, 8 Placebo tablets over a 4hr schedule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylene Blue MMX®
  Other Names: Investigational Product: Methylene Blue MMX® modified release tablets; Active Ingredient: Methylene Blue
  Arms: Methylene Blue MMX® 100mg; Methylene Blue MMX® 200mg
Drug: Placebo — Sugar pill manufactured to mimic Methylene Blue MMX® tablet.
  Arms: Methylene Blue MMX® 100mg; Placebo

SUMMARY:
Evaluation of the histologically proven adenoma and carcinoma detection rate in patients undergoing a full colonoscopy with and without mucosal contrast enhancement, obtained with 200 mg of Methylene Blue MMX® tablets.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, aged between 50 and 75.
* Outpatients scheduled for screening or surveillance colonoscopy for polyps or colorectal cancer )
* Able to comprehend the full nature and purpose of the study, including possible risks and side effects.
* Able to co-operate with the investigator and to comply with the requirements of the entire study.
* Signed written informed consent prior to inclusion in the study.

Exclusion Criteria:

* Patients at high risk of colorectal cancer e.g. ulcerative colitis
* Previous medical history of, or suspected hypersensitivity to, the Methylene Blue and/or formulations' ingredients.
* Previous medical history of, or suspected hypersensitivity to, the PEG based bowel cleansing preparation and/or bowel cleansing formulations' ingredients.
* Previous medical history of gastrointestinal obstruction or perforation, toxic megacolon, major colonic resection, severe diverticulitis, heart failure (Class III or IV), serious cardiovascular disease, ulcerative colitis or Crohn's disease.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1249 (Actual)
Dates: Start 2013-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Repici, MD, Principal Investigator — Co-ordinating Investigator EU; Michael Wallace, MD, Principal Investigator — Co-ordinating Investigator US
Locations (19):
- United States (7):
  - Dr Michelle Young, Phoenix, Arizona
  - Dr Francesco Ramirez, Scottsdale, Arizona
  - Dr David Gatof, Lafayette, Colorado
  - Dr Michael Wallace, Jacksonville, Florida
  - Dr Prateek Sharma, Kansas City, Kansas
  - Dr Marcia Canto, Baltimore, Maryland
  - Dr David Bruining, Rochester, Minnesota
- Dr Raf Bisschop, Leuven, Belgium
- Dr Norman Marcon, Toronto, Ontario, Canada
- Dr Ralf Kiesslich, Wiesbaden, Germany
- Italy (3):
  - Dr Renato Cannizzaro, Aviano
  - Dr Cesare Hassan, Rome
  - Dr Alessandro Repici, Rozzano
- Dr Limas Kupcinskas, Kaunas, Lithuania
- Netherlands (3):
  - Dr Evelien Dekker, Amsterdam
  - Dr Manoon Spander, Rotterdam
  - Dr Peter Siersema, Utrecht
- United Kingdom (2):
  - Dr James East, Oxford
  - Dr Matthew Rutter, Stockton-on-Tees

REFERENCES:
- [Derived] Repici A, Wallace MB, East JE, Sharma P, Ramirez FC, Bruining DH, Young M, Gatof D, Irene Mimi Canto M, Marcon N, Cannizzaro R, Kiesslich R, Rutter M, Dekker E, Siersema PD, Spaander M, Kupcinskas L, Jonaitis L, Bisschops R, Radaelli F, Bhandari P, Wilson A, Early D, Gupta N, Vieth M, Lauwers GY, Rossini M, Hassan C. Efficacy of Per-oral Methylene Blue Formulation for Screening Colonoscopy. Gastroenterology. 2019 Jun;156(8):2198-2207.e1. doi: 10.1053/j.gastro.2019.02.001. Epub 2019 Feb 10. PMID 30742834

RESULTS

PARTICIPANT FLOW:
Groups:
- Methylene Blue MMX® 200mg: Oral dose, 8 Methylene Blue MMX® tablets over a 4hr schedule
  Methylene Blue MMX®
- Methylene Blue MMX® 100mg: Oral dose, 4 Methylene Blue MMX® tablets and 4 Placebo tablets over a 4hr schedule
  Methylene Blue MMX®
  Placebo: Sugar pill manufactured to mimic Methylene Blue MMX® tablet.
Period: Overall Study
Arm/Group | Methylene Blue MMX® 200mg | Methylene Blue MMX® 100mg | Placebo
Started | 504 | 247 | 498
Completed | 470 | 232 | 464
Not Completed | 34 | 15 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methylene Blue MMX® 200mg | Methylene Blue MMX® 100mg | Placebo | Total
Number analyzed (Participants) | 504 | 247 | 498 | 1249
Age, Categorical [Count of Participants; unit: Participants] — Population: ITT=1249, FAS=1205
  Participants
    number analyzed (Participants) | 485 | 241 | 479 | 1205
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 313 | 163 | 298 | 774
    >=65 years | 172 | 78 | 181 | 431
Sex: Female, Male [Count of Participants; unit: Participants] — Population: ITT=1249 FAS=1205
  Participants
    number analyzed (Participants) | 485 | 241 | 479 | 1205
    Female | 191 | 103 | 184 | 478
    Male | 294 | 138 | 295 | 727

OUTCOME MEASURES:

1. Primary Outcome: To Assess the Detection Efficacy of Chromoendoscopy Performed With 200mg Methylene Blue MMX® 25 mg Tablets Versus Placebo Tablets (White Light Endoscopy) in Terms of the Proportion of Subjects With at Least One Histologically Proven Adenoma or Carcinoma.
Description: Adenoma Detection Rate
Time Frame: +7 days
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Methylene Blue MMX® 200mg | Methylene Blue MMX® 100mg | Placebo
Number analyzed (Participants) | 485 | 241 | 479
percentage of participants | 56.3 | 51.5 | 47.8

ADVERSE EVENTS:
Arm/Group | Methylene Blue MMX® 200mg | Methylene Blue MMX® 100mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/485 | 1/241 | 0/479
Other Adverse Events (participants affected / at risk) | 234/488 | 102/241 | 7/479
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methylene Blue MMX® 200mg (N=485) | Methylene Blue MMX® 100mg (N=241) | Placebo (N=479)
viral bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methylene Blue MMX® 200mg (N=488) | Methylene Blue MMX® 100mg (N=241) | Placebo (N=479)
faeces discoloured (Gastrointestinal disorders) | 95 (95) | 43 (43) | 0 (0)
chromaturia (Renal and urinary disorders) | 234 (234) | 102 (102) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications to be reviewed by sponsor prior to submission.